CLINICAL TRIAL: NCT01055119
Title: Effect of Supplementation With Long Chain Polyunsaturated Fatty Acids on Behavior and Cognition in Children With Attention Deficit Hyperactivity Disorder
Brief Title: Effect of Long Chain Polyunsaturated Fatty Acids on Behavior and Cognition in Children With Attention Deficit Hyperactivity Disorder
Acronym: EFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Katharina Widenhorn-Mueller, Katharina Widenhorn-Mueller, PhD, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: ADHD PUFA 2009
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 fatty acids (Active Comparator)
  Interventions: Dietary Supplement: Omega-3 fatty acids
- Olive oil (Placebo Comparator)
  Interventions: Dietary Supplement: Omega-3 fatty acids

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acids — duration: 4 month

SUMMARY:
The study investigates whether eicosapentaenoic/docosahexaenoic acid supplementation affects behavior and cognition in children with attention deficit hyperactivity disorder.

ELIGIBILITY:
Inclusion Criteria:

* ADHD diagnosis
* Age 9-12y
* Native German speaker

Exclusion Criteria:

* Allergy against fish and fish products
* IQ below 85
* Objections against pork gelatine

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2009-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Behavior, Cognition | Before intervention and 16 weeks after start of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Bode Harald, MD, Principal Investigator — Sozialpädiatrisches Zentrum und Kinderneurologie Universitätsklinik für Kinder- und Jugendmedizin, Ulm University
Locations (2):
- Germany (2):
  - Klinik fuer Psychiatrie und Psychotherapie III, Ulm, Baden-Wurttemberg
  - Universitaet Ulm Klinik fuer Psychiatrie und Psychotherapie III, Ulm